CLINICAL TRIAL: NCT02171923
Title: Medial Prefrontal Cortex and Vulnerability for Depression
Brief Title: Multicenter Comparative Study of the Activity of the Medial Prefrontal Cortex in Vulnerability to Depression
Acronym: CORVAD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110139
Record Dates: First submitted 2013-09-17; First posted 2014-06-24 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Major Depression
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Remitted depressed patients: Formerly depressed patients in remission for 6 months or more
- healthy controls: healthy subjects with no history of mental disorders

SUMMARY:
To examine whether the medial prefrontal cortex displays an increased activity during self-referential processing among remitted depressed patients compared to healthy controls

ELIGIBILITY:
Inclusion criteria (patients)

* History of at least one major depressive episode
* In clinical remission for at least 6 months (BDI-21 ≤ 10 & Montgomery and Asberg Depression Rating Scale ≤ 7)
* Aged 20-65

Exclusion criteria :

* first depressive episode after the age of 59
* last episode treated by cognitive behavior therapy
* currently receiving a antipsychotic or mood-stabilizing drug
* personal history of: major depressive episode with psychotic features, other axis-I disorder (except generalized anxiety disorder), substance-related disorder (except nicotine dependence), bipolar disorder
* first-degree familial history of bipolar disorder
* cognitive impairment due to another central nervous system disease
* contra-indication to MRI
* pregnancy
* refusal to be informed of abnormal findings during the MRI

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Formerly depressed patients and healthy controls matched for age and sex
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
BOLD signal in the medial prefrontal cortex | 18 month
  Each subject will have a standardized psychometric assessment (BDI-21, MADRS, STAI, RRS) in a Siemens 3T Trio for collecting voxel BOLD signal (Blood-Oxygen-Level Dependent). For each subject and each voxel, a coefficient beta relative activation will be obtained with a general linear model using the timing of presentation of stimuli and the expected signal to model the measured hemodynamic BOLD response. A main effect of condition (personal versus general) will be sought to determine the peak activation within the dorsal CMPF (defined region of interest using the Pickatlas software). The primary endpoint will be the beta coefficient on the level of activation of a sphere 10 mm in diameter centered on the peak.

SECONDARY OUTCOMES:
depression relapse | 1 year
  The presence (MINI) and intensity (BDI) for possible depressive relapse will be sought from the attending psychiatrist and during telephone interviews at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Lemogne, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- URC - HEGP, 20 rue Leblanc, Paris, France

REFERENCES:
- [Background] Lemogne C, Delaveau P, Freton M, Guionnet S, Fossati P. Medial prefrontal cortex and the self in major depression. J Affect Disord. 2012 Jan;136(1-2):e1-e11. doi: 10.1016/j.jad.2010.11.034. Epub 2010 Dec 23. PMID 21185083